CLINICAL TRIAL: NCT03584555
Title: Comparison of Clinical Outcomes of Small-incision Lenticule Extraction (SMILE) Between Different Cap Thickness.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2017-0063
Record Dates: First submitted 2018-06-19; First posted 2018-07-12 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Myopia
Keywords: Small incision lenticule extraction; Cap thickness
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: Enrollment period : 24 months after IRB approval Methods: The subjects are randomly divided into two groups. One group underwent SMILE surgery using 120 μm cap thickness, and the other group underwent SMILE surgery using 140 μm cap thickness. Before surgery, all patients underwent a detailed ophthalmological examination that included evaluation of logarithm of the minimum angle of resolution (logMAR) uncorrected-distance visual acuity (UDVA) and CDVA, manifest refraction, slit-lamp examination (Haag-Streit, Köniz, Switzerland), keratometry, and Scheimpflug-based corneal topography (Pentacam HR, Oculus). Dynamic corneal response (DCR) parameters were examined using Corvis ST. Corneal wavefront aberrations were measured using Keratron Scout (Optikon 2000, Rome, Italy). All examinations were repeated at 1, 3, and 6 months after surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 120 μm group (Active Comparator): The subjects underwent SMILE using 120 μm cap.
  Interventions: Procedure: SMILE using 120μm cap thickness
- 140 μm group (Active Comparator): The subjects underwent SMILE using 140 μm cap.
  Interventions: Procedure: SMILE using 140μm cap thickness

INTERVENTIONS:
Procedure: SMILE using 120μm cap thickness — The surgery was performed with standardized techniques with triple centration technique using the 500-KHz VisuMax system (Carl Zeiss Meditec AG, Jena, Germany). The superior cap depth was set as 120 or 140 µm, and the length of the side cut was set to 2 mm. Once the anterior (upper) and posterior (lower) planes of the lenticule were defined, the anterior and posterior interfaces were dissected using a micropetala with a blunt circular tip and extracted with midforceps. The integrity of the lenticule was assessed subsequently.
  Arms: 120 μm group
Procedure: SMILE using 140μm cap thickness — The surgery was performed with standardized techniques with triple centration technique using the 500-KHz VisuMax system (Carl Zeiss Meditec AG, Jena, Germany). The superior cap depth was set as 120 or 140 µm, and the length of the side cut was set to 2 mm. Once the anterior (upper) and posterior (lower) planes of the lenticule were defined, the anterior and posterior interfaces were dissected using a micropetala with a blunt circular tip and extracted with midforceps. The integrity of the lenticule was assessed subsequently.
  Arms: 140 μm group

SUMMARY:
In the past two decades, the femtosecond laser (FSL) technology has been introduced in the corneal refractive surgery filed, and brought a remarkable innovation. It can make tissue dissection through photodisruption and plasma cavitation. Initially, the FSL was used predominantly to make a corneal flap when performing laser in situ keratomileusis (LASIK), which is followed by stromal ablation using excimer laser. A new surgical technique called femtosecond lenticule extraction (FLEx) has been developed that uses only FSL to dissect two interfaces to create refractive lenticule and then remove it, which is very similar with LASIK. Small incision lenticule extraction (SMILE) which is the advanced form of all-in-one FSL refractive technique does not make a corneal flap rather make small incision where the separated refractive lenticule is removed through, and the upper part of the corneal tissue is called cap. Since the clinical outcomes of SMILE were firstly published in 2011, SMILE has been widely used for correction of myopia or myopic astigmatism worldwide. SMILE provides excellent visual outcomes and has advantages including a lesser decrease in corneal sensitivity and absence of flap related complications compared to LASIK.

Because corneal ectasia after refractive surgery is the one of most terrifying complication, corneal biomechanics has been drawn interests to many researchers and clinicians. Theoretically, SMILE may preserve corneal biomechanics better than LASIK, because the anterior stroma which is stiffer than the posterior stroma remains intact in SMILE. However, there are some controversies, because previous studies investigating corneal biomechanics have been reported inconsistent outcomes, although SMILE has been reported equal to or better than LASIK. Weakening of corneal biomechanics and iatrogenic corneal ectasia have also been reported after SMILE. In addition, because the tensile strength of cornea gradually decreases as it goes backwards, creating deeper refractive lenticule may result in stronger cornea by preserving more of anterior lamellae of the cornea. But on the contrary, leaving sufficient residual stromal bed has been known to be important in preventing iatrogenic corneal ectasia, hence creating thin cap may be effective and desirable. Although many researches have been investigated the difference in biomechanical response between SMILE and LASIK, there are few studies evaluating the dependence of cap thickness on postoperative biomechanical strength after SMILE. El-Massry et al. reported that the thicker cap thickness showed higher postoperative corneal hysteresis (CH) and corneal resistance factor (CRF) with Ocular Response Analyzer (ORA; Reichert Ophthalmic Instruments, Depew, NY) which may not be optimal for a clear description of the viscosity and elasticity of the cornea,3 ; however, other studies have been presented that there is no significant difference of corneal biomechanics with cap thickness. There is no comparative human study using Corvis ST (Oculus, Wetzlar, Germany) despite presence of the study using Corvis ST in rabbit eyes. Furthermore, no prospective study with large number of subjects has been performed to date.

ELIGIBILITY:
Inclusion Criteria:

1. age of 20 years or older.
2. Myopia
3. Who is willing to get SMILE surgery

Exclusion Criteria:

1. severe ocular surface disease
2. any corneal disease, cataract, glaucoma, macular disease, or previous history of intraocular or corneal surgery
3. Patients with suspicion of keratoconus on corneal topography

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2017-03-18 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
Uncorrected Distance Vision Acuity | from preoperative to postoperative 6 months
  Uncorrected Distance Vision Acuity in logMAR scale will be compared between the two groups at each time point.
Corrected Distance vision Acuity | from preoperative to postoperative 6 months
  Corrected Distance Vision Acuity in logMAR scale will be compared between the two groups at each time point.

SECONDARY OUTCOMES:
1.Total higher order aberration at each time point between the two groups. | from preoperative to postoperative 6 months
  Total higher order aberrations, spherical aberrations, and coma aberrations are examined using Keratron Scout (Optikon 2000, Rome, Italy). The unit of those is "μm".
  1,2. Total higher order aberrations at each time point and change from baseline at each time point will be compared between the two groups.
2.Total higher order aberration changes from baseline at each postoperative time point between the two groups. | from preoperative to postoperative 6 months
  Total higher order aberrations, spherical aberrations, and coma aberrations are examined using Keratron Scout (Optikon 2000, Rome, Italy). The unit of those is "μm".
  1,2. Total higher order aberrations at each time point and change from baseline at each time point will be compared between the two groups.
3.Spherical aberration at each time point between the two groups. | from preoperative to postoperative 6 months
  3,4. Spherical aberrations at each time point and change from baseline at each time point will be compared between the two groups.
4.Spherical aberration changes from baseline at each postoperative time point between the two groups. | from preoperative to postoperative 6 months
  3,4. Spherical aberrations at each time point and change from baseline at each time point will be compared between the two groups.
5.Coma aberration at each time point between the two groups. | from preoperative to postoperative 6 months
  5,6. Coma aberrations at each time point and change from baseline at each time point will be compared between the two groups.
  Corneal biomechanics including deformation amplitude ratio (DA ratio), and stiffness parameter at first applanation (SP-A1) is examined using Corvis ST (Oculus, Wetzlar, Germany). The unit of SP-A1 is "mm Hg/mm", and DA ratio is unitless.
6.Coma aberration changes from baseline at each postoperative time point between the two groups. | from preoperative to postoperative 6 months
  5,6. Coma aberrations at each time point and change from baseline at each time point will be compared between the two groups.
  Corneal biomechanics including deformation amplitude ratio (DA ratio), and stiffness parameter at first applanation (SP-A1) is examined using Corvis ST (Oculus, Wetzlar, Germany). The unit of SP-A1 is "mm Hg/mm", and DA ratio is unitless.
7.Deformation amplitude ratio (DA ratio) at each time point between the two groups. | from preoperative to postoperative 6 months
  7,8 DA ratio at each time point and change from baseline at each time point will be compared between the two groups.
8.DA ratio changes from baseline at each postoperative time point between the two groups. | from preoperative to postoperative 6 months
  7,8 DA ratio at each time point and change from baseline at each time point will be compared between the two groups.
9.Stiffness parameter at first applanation (SP-A1) at each time point between the two groups. | from preoperative to postoperative 6 months
  9,10 SP-A1 at each time point and change from baseline at each time point will be compared between the two groups.
10.SP-A1 changes from baseline at each postoperative time point between the two groups. | from preoperative to postoperative 6 months
  9,10 SP-A1 at each time point and change from baseline at each time point will be compared between the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Yonsei Univeristy College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Damgaard IB, Ivarsen A, Hjortdal J. Refractive Correction and Biomechanical Strength Following SMILE With a 110- or 160-mum Cap Thickness, Evaluated Ex Vivo by Inflation Test. Invest Ophthalmol Vis Sci. 2018 Apr 1;59(5):1836-1843. doi: 10.1167/iovs.17-23675. PMID 29610851
- [Background] Fernandez J, Rodriguez-Vallejo M, Martinez J, Tauste A, Pinero DP. Corneal biomechanics after laser refractive surgery: Unmasking differences between techniques. J Cataract Refract Surg. 2018 Mar;44(3):390-398. doi: 10.1016/j.jcrs.2017.10.054. Epub 2018 Mar 31. PMID 29615281
- [Background] Weng S, Liu M, Yang X, Liu F, Zhou Y, Lin H, Liu Q. Evaluation of Human Corneal Lenticule Quality After SMILE With Different Cap Thicknesses Using Scanning Electron Microscopy. Cornea. 2018 Jan;37(1):59-65. doi: 10.1097/ICO.0000000000001404. PMID 29053560
- [Background] He M, Wang W, Ding H, Zhong X. Comparison of Two Cap Thickness in Small Incision Lenticule Extraction: 100mum versus 160mum. PLoS One. 2016 Sep 21;11(9):e0163259. doi: 10.1371/journal.pone.0163259. eCollection 2016. PMID 27655417
- [Background] Liu M, Zhou Y, Wu X, Ye T, Liu Q. Comparison of 120- and 140-mum SMILE Cap Thickness Results in Eyes With Thick Corneas. Cornea. 2016 Oct;35(10):1308-14. doi: 10.1097/ICO.0000000000000924. PMID 27467038
- [Background] El-Massry AA, Goweida MB, Shama Ael-S, Elkhawaga MH, Abdalla MF. Contralateral Eye Comparison Between Femtosecond Small Incision Intrastromal Lenticule Extraction at Depths of 100 and 160 mum. Cornea. 2015 Oct;34(10):1272-5. doi: 10.1097/ICO.0000000000000571. PMID 26266430